CLINICAL TRIAL: NCT00952120
Title: Comparison of Two Methods of Securing Skin Grafts Using Negative Pressure Wound Therapy: VAC and GSUC
Brief Title: Comparison of Two Methods of Securing Skin Grafts Using Negative Pressure Wound Therapy: Vacuum Assisted Closure (VAC) and Gauze Suction (GSUC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16863B
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Results first posted 2015-09-24 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-08

CONDITIONS: Wound Healing
Keywords: Wound healing; Negative pressure wound therapy; Skin graft

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSUC (Experimental): Gauze-based wall suction negative pressure wound therapy for 4-5 days
  Interventions: Device: GSUC
- Vacuum-assisted closure (Active Comparator): Vacuum-assisted closure (VAC) negative pressure wound therapy using commercially available device (KCI, Inc) for 4-5 days
  Interventions: Device: VAC

INTERVENTIONS:
Device: GSUC — Gauze-based wall suction negative pressure wound therapy
  Arms: GSUC
Device: VAC — Commercially available Wound VAC negative pressure wound therapy device (KCI, Inc.)
  Arms: Vacuum-assisted closure

SUMMARY:
The purpose of this study is to compare how well two methods (VAC and G-SUC) of securing skin grafts using negative pressure wound therapy work. Negative pressure wound therapy is a commonly used method of applying suction on wounds to remove fluid from wound and to promote healing. The VAC system is widely used and consists of a foam dressing and a portable computerized suction pump. The G-SUC method uses commonly available dressing supplies attached to vacuum (suction) pump located on the wall above a hospital bed. The investigators have frequently used both methods over the past 10 years and have not observed any specific negative side effects of either.

DETAILED DESCRIPTION:
STUDY DESIGN: A prospective, randomized study will be conducted. The investigators expect the duration of data collection to be 2 years.

1. PATIENT SELECTION

   Adult patients of any sex, hospitalized at the University of Chicago Medical Center, requiring split thickness skin autografts with wounds that are amenable to placement of an occlusive dressing for negative pressure therapy will be eligible to participate in the study. If both the patient and the primary treating surgeon agree to participate, they will receive informed consent. Pregnant women, children under 18 years of age and other patients who are "vulnerable" as defined by the Institutional Review Board will not be eligible for the study.
2. STUDY PROCEDURE

Preoperative Procedures:

Patients with wounds requiring skin grafting will enter the trial upon consent of the patient and the preoperative decision by the surgeon to secure the skin graft with negative pressure therapy. Upon entry, the primary physical therapist will be immediately informed of a study participant and will place either the G-SUC or VAC dressing at the conclusion of the operation. The randomization scheme will be prepared by the study statistician using computer generated random numbers. The surgeon will be blinded to the treatment modality until the primary physical therapist places the randomized therapy.

Intraoperative Procedures:

Wounds will undergo debridement using standard techniques to a healthy, viable wound bed. Split thickness skin grafts harvested from the patient will be obtained between 0.008-0.010 inches using an electric dermatome. In addition to standard methods of achieving hemostasis, Tisseel (Baxter, Deerfield, IL) will be used as an adjunct for the preparation of the wound bed. All grafts will be secured with N-Terface Interpositional Material (Winfield Laboratories, Richardson, TX) and a single layer of Acticoat (Smith and Nephew, Quebec, Canada).

Patients with skin grafts undergoing VAC therapy will be managed with continuous negative pressure delivered by the computerized VAC suction unit at 75-125 mm Hg. The suction will be applied to a standard open cell VAC foam dressing supplied by KCI, Inc and sealed with an occlusive cover.

Patients with skin grafts undergoing G-SUC therapy will be managed with negative pressure delivered by low continuous wall suction at 75-80 mm Hg. The suction will be applied to standard gauze dressing and sealed with an occlusive cover.

Postoperative Procedures:

Patients on either therapy will remain on continuous negative pressure therapy from the conclusion of their surgery until dressing takedown. Patients undergoing VAC therapy will be transported with the computerized VAC suction unit. Maintenance of negative pressure during transport of patients undergoing G-SUC therapy will be accomplished by clamping the connection tubing with hemostats prior to disconnection to wall suction units.

All dressings will be discontinued on post operative day #4 or 5 and graft take will be assessed with two methods in the following manner:

1. Areas of non-take will be clearly marked with a pen by a researcher blinded to the treatment modality
2. Images of the graft with a ruler for scale will be taken by a digital camera
3. The entire graft area will be determined in pixels
4. The areas of non-take will be determined in pixels
5. The percentage of non-take will then be calculated
6. The areas will also be measured and recorded

Image analysis will be conducted by a researcher blinded to the treatment modality. Wound size will also be calculated as per Xakellis & Frantz method (1997): wound surface area = length x width x 0.783.

If a G-SUC or VAC dressing cannot be maintained because of either persistent fluid or suction leaks, the attending physical therapist will attempt to reinforce the dressing. If after 2 attempts per 24-hour period, the dressing still cannot be maintained, that patient will be considered to have failed negative pressure wound therapy. Patients who fall into this category will be able to crossover into the other treatment arm, but additional data regarding their treatment will not considered in the results of the study.

The cost of VAC rental, supplies and time performing dressing changes will be recorded for the duration of negative pressure wound therapy for each patient.

The attending physical therapist will collect and maintain the database.

Wound Specific Procedures:

Upper Extremity. All skin grafts on mobile structures, such as those crossing joints or directly on muscle, will be splinted to prevent shear. Otherwise, patients will be allowed to move about ad lib.

Lower Extremity. All skin grafts on mobile structures, such as those crossing joints or directly on muscle, will be splinted to prevent shear. Patients will remain on bedrest with leg elevation to prevent lower extremity edema until negative pressure therapy is discontinued.

Chest, Abdomen, Back, Head, Neck. Mobility will be allowed ad lib.

Perineum. Patients will remain on bedrest until discontinuation of negative pressure therapy to prevent shear.

3. STUDY RECORDS

Completed case report forms will be confidential and kept in a secured file by the principal investigator.

4. RISKS & BENEFITS TO PATIENTS

The investigators are not aware that there are specific risks associated with negative pressure wound therapy, and the technique has not been associated with specific adverse outcomes at our hospital or in the published literature. Negative pressure wound therapy allows for more rapid and reliable wound healing for many patients. Data from this study may help us to expand the indications for negative pressure wound therapy.

There will be no payment to the subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of any sex, hospitalized at the University of Chicago Medical Center, requiring split thickness skin autografts with wounds that are amenable to placement of an occlusive dressing for negative pressure therapy will be eligible to participate in the study

Exclusion Criteria:

* Pregnant women, children under 18 years of age and other patients who are "vulnerable" as defined by the Institutional Review Board will not be eligible for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-05; Primary Completion 2011-12 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Gottlieb, MD, Principal Investigator — University of Chicago, Section of Plastic and Reconstructive Surgery
Locations (1):
- University of Chicago Medical Center, Section of Plastic and Reconstructive Surgery, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 104 unique patients were enrolled with a total of 157 wounds (80 of the wounds received GSUC and 77 of the wounds received vacuum-assisted closure).
Groups:
- GSUC: Continuous negative pressure therapy from the conclusion of the surgery until dressings were taken down on postoperative day 4 or 5. The negative pressure was delivered by low continuous wall suction at 50 to 125 mmHg via a red rubber catheter placed within standardized gauze dressing moistening with sterile saline and sealed with Ioban occlusive dressing.
- Vacuum-assisted Closure: Continuous negative pressure therapy from the conclusion of the surgery until dressings were taken down on postoperative day 4 or 5. The negative pressure was delivered by the VAC suction unit at 30 to 125 mmHg through a open cell VAC foam dressing sealed with an occlusive cover.
- GSUC and Vacuum-assisted Closure: These patients had multiple wounds and some of their wounds received GSUC therapy and some of their wounds received VAC.
Period: Overall Study
Arm/Group | GSUC | Vacuum-assisted Closure | GSUC and Vacuum-assisted Closure
Started | 52 | 47 | 5
Completed | 52 | 47 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: 104 unique patients were enrolled with a total of 157 wounds (80 of the wounds received GSUC and 77 of the wounds received vacuum-assisted closure).
Groups:
- Total: Total of all reporting groups
Arm/Group | GSUC | Vacuum-assisted Closure | GSUC and Vacuum-assisted Closure | Total
Number analyzed (Participants) | 52 | 47 | 5 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (16.5) | 50.1 (16.4) | 51.8 (20.7) | 51.4 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 2 | 52
  Male | 27 | 22 | 3 | 52
Region of Enrollment [Number; unit: participants]
  United States | 52 | 47 | 5 | 104

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Wounds With Complete Skin Graft Take
Description: For each wound, the percentage of the skin graft that took by Day 4 or 5 was calculated. Complete take is defined as 100% take or skin graft incorporation.
Time Frame: Day 4 or 5
Population: Some patients had multiple wounds that required skin grafting. Wounds were the unit of analysis, so a participant with multiple wounds could be in both treatment groups which is why the total number of participants adds to more than the number of unique participants enrolled in the study (and included in the participant flow and baseline tables).
Measure: Number; unit: percentage of wounds
Units Other Than Participants: wounds
Groups:
- Vacuum-assisted Closure: VAC negative pressure wound therapy using commercially available device (KCI, Inc) for 4-5 days
  VAC: Commercially available Wound VAC negative pressure wound therapy device (KCI, Inc.)
Arm/Group | GSUC | Vacuum-assisted Closure
Number analyzed (Participants) | 57 | 53
Number analyzed (wounds) | 80 | 77
percentage of wounds | 80 | 78
Statistical Analysis 1: Comparison: GSUC vs Vacuum-assisted Closure; Test type: Superiority or Other; p = 0.80, Regression, Logistic; robust standard errors were used to account for the multiple observations per patient

2. Secondary Outcome: Percentage of Wounds With Total Skin Graft Loss
Description: For each wound, whether there was total skin graft loss by Day 4 or 5 was determined.
Time Frame: Day 4 or 5
Population: as for outcome 1
Measure: Number; unit: percentage of wounds
Units Other Than Participants: wounds
Arm/Group | GSUC | Vacuum-assisted Closure
Number analyzed (Participants) | 57 | 53
Number analyzed (wounds) | 80 | 77
percentage of wounds | 3.8 | 1.3

ADVERSE EVENTS:
Time Frame: 4 or 5 days
Description: Some patients had multiple wounds that required skin grafting. Wounds were the unit of analysis, so a participant with multiple wounds could be in both treatment groups which is why the total number of participants adds to more than the number of unique participants enrolled in the study (and included in the participant flow and baseline tables)
Arm/Group | GSUC | Vacuum-assisted Closure
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/53
Other Adverse Events (participants affected / at risk) | 0/57 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes